CLINICAL TRIAL: NCT05401929
Title: Imaging the Effects of Intermittent Thetaburst Stimulation on Cannabis Self-Administration in Heavy Cannabis Users
Brief Title: Transcranial Magnetic Brain Stimulation to Reduce Cannabis Use in Heavy Cannabis Users
Acronym: iCURE
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: June 2023 NYSPI began safety review of all human subjects research, so ongoing studies paused June 12. DHHS OHRP also issued FWA restriction on NYSPI research that included pause of human research on June 23. Research will resume upon review.
Sponsor: Duke University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00118090; K01DA050691 (NIH)
Record Dates: First submitted 2022-05-27; First posted 2022-06-02 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Cannabis
Keywords: cannabis; transcranial magnetic stimulation; repetitive transcranial magnetic stimulation; intermittent theta burst stimulation; functional magnetic resonance imaging; functional neuroimaging; functional brain imaging; marijuana; cannabis smoking; marijuana smoking; recreational marijuana use; stroop task; attentional bias; drug cue reactivity; intervention; treatment; double blind; sham; sham controlled; ecological momentary assessment; randomized controlled clinical trials; randomized clinical trials; neuronavigation; personalized cortical targeting; biomarker development; brain mapping; neuroendophenotypes; neurobiomarkers; accelerated; functional connectivity; network; fmri
MeSH Terms: conditions — Marijuana Abuse; Marijuana Smoking; Marijuana Use | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active (Experimental)
  Interventions: Device: iTBS
- Sham (Sham Comparator)
  Interventions: Device: iTBS

INTERVENTIONS:
Device: iTBS — Sixty trains of active intermittent thetaburst stimulation (iTBS) (1 train = 10 sec of 2 sec ON, 8 sec OFF; 3-pulse bursts at 5 Hz; 15 pulses/sec [30 pulses/train]; 60 trains/session; 1,800 pulses/session) using neuronavigation-guided cortical targeting to the left dorsolateral prefrontal cortex location using figure-of-8 TMS coils.
  Other Names: Repetitive transcranial magnetic stimulation; Patterned repetitive transcranial magnetic stimulation; rTMS; intermittent thetaburst stimulation; Intermittent theta burst stimulation; Intermittent theta-burst stimulation; accelerated; accelerated iTBS; accelerated rTMS
  Arms: Active
Device: iTBS — Sixty trains of sham intermittent thetaburst stimulation (iTBS) (1 train = 10 sec of 2 sec ON, 8 sec OFF; 3-pulse bursts at 5 Hz; 15 pulses/sec [30 pulses/train]; 60 trains/session; 1,800 pulses/session) using neuronavigation-guided cortical targeting to the left dorsolateral prefrontal cortex location using figure-of-8 TMS coils.
  Arms: Sham

SUMMARY:
The growing legalization of cannabis across the U.S. is associated with increases in cannabis use, and accordingly, an increase in the number of individuals with cannabis use problems, including cannabis use disorder (CUD). While there are several medications being investigated as treatment options for CUD, none have been FDA-approved, and there is limited efficacy of traditional behavioral therapy approaches for this population. Consequently, there is a pressing need for the development of new treatments, including approaches that specifically target the brain areas associated with problematic cannabis use behaviors. Elevated attention to drug cues is one of the primary causes of relapse in heavy cannabis users. Preliminary data suggests that repetitive transcranial magnetic stimulation (rTMS), a non-invasive form of brain stimulation, may be a novel brain-based tool to decrease heightened attention to drug cues in people with CUD. Building on prior data, the primary goal of this study is to evaluate the feasibility and effectiveness of TMS as a tool to decrease attention to drug cues and reduce cannabis use.

In this study, fifty (50) treatment-seeking, near-daily cannabis users will be recruited to receive either active or sham (placebo) repetitive TMS (rTMS). Participants will complete a total of 25 treatment sessions, delivered as five sessions per day across five days, with sessions flexibly scheduled over a two-week period. Measures of cannabis use and brain activity will be collected before and after treatment using real-time self-report assessments and functional magnetic resonance imaging (fMRI), respectively. Specifically, cannabis use will be assessed in participants' everyday environments using brief text-message surveys during a two-week baseline period, the two-week treatment period, and a four-week follow-up period.

The study aims to determine whether active rTMS reduces brain activity in response to cannabis cues, decreases automatic attention to cannabis cues, and leads to meaningful reductions in cannabis use compared to sham treatment.

DETAILED DESCRIPTION:
The expanding legalization of cannabis across the U.S. is associated with increases in cannabis use and, accordingly, an increase in the number of individuals with cannabis use disorder (CUD). One key predictor of relapse is elevated attentional bias to drug cues, coupled with attenuated cognitive control in the presence of those cues. Attentional bias to drug cues is associated with increased activity in the Salience Network (SN), including the anterior cingulate cortex and bilateral anterior insula, as well as reduced activity in the dorsolateral prefrontal cortex (DLPFC) and broader cognitive control circuitry during exposure to cannabis cues.

Our prior data demonstrate that neural responses to drug cues can be reduced by attenuating ventromedial prefrontal cortex (VMPFC) and reward circuitry using inhibitory repetitive transcranial magnetic stimulation (rTMS) (Strategy 1). An alternative approach, however, may be to enhance activity in the DLPFC and cognitive control circuitry, which may also reduce neural reactivity to drug cues by inversely regulating SN cue hyper-reactivity (Strategy 2, the focus of this K01). Through the research and training plan outlined in this K01 proposal, I seek to evaluate the ability of left DLPFC-targeted rTMS to attenuate SN drug cue reactivity and attentional bias, and to reduce cannabis use. This will be accomplished by applying accelerated intermittent theta burst stimulation (aiTBS), a novel patterned excitatory form of rTMS, to the L DLPFC in heavy cannabis users.

GOAL. The primary objectives of this K01 research project are to:

1. determine whether L DLPFC aiTBS decreases cannabis use using real-time data collected in the natural environment;
2. determine whether aiTBS-induced changes in cannabis use are associated with changes in Salience Network drug cue reactivity; and
3. assess whether L DLPFC aiTBS is feasible, tolerable, and safe relative to sham stimulation.

DESIGN. Fifty (50) treatment-seeking, heavy (near-daily) cannabis users will be randomized to receive either active or sham aiTBS targeting the L DLPFC. Participants will complete a total of 25 treatment sessions, delivered as five sessions per day (50-min inter-session interval) across five treatment days, with visits flexibly scheduled over a two-week period. Cannabis use data will be collected throughout the study, and functional magnetic resonance imaging (fMRI) data will be collected before and after aiTBS treatment, as well as following a 4-week follow-up period.

Cannabis use in the natural environment will be assessed using Ecological Momentary Assessment (EMA) during a two-week baseline (pre-treatment) period, a two-week treatment period, and a four-week follow-up period. Frequency of use (days per week) and quantity of use (average grams per use day) will be captured via EMA and corroborated during the four follow-up visits using Timeline Followback (TLFB) interviews and urine toxicology to assess cannabis and other substance use and to monitor for adverse events.

We will test the hypotheses that active aiTBS will reduce neural reactivity to cannabis cues (Aim 2), reduce cannabis use frequency and/or quantity (Aim 1), and demonstrate non-inferior feasibility, tolerability, and safety compared to sham stimulation (Safety Aim).

Over the two-year recruitment period, this project will generate a critical dataset to advance brain stimulation treatment development for CUD. In addition, these data will support a subsequent R01 application aimed at extending this line of treatment development research. Finally, this project will provide essential training in human behavioral pharmacology and clinical trial research design and analysis, supporting my progression toward independence as an interdisciplinary addiction neuroscientist.

ELIGIBILITY:
Inclusion Criteria:

* Males/non-pregnant females, 18-65 years old
* Current cannabis user
* Able to perform all study procedures

Exclusion Criteria:

* Regular use of other illicit drugs
* If medical history, physical and psychiatric examination, or laboratory tests performed during the screening process reveal any significant illness that the study physician deems contraindicated for study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Frequency of cannabis use | Two-week Pre-treatment/Baseline phase (Days 1-14), Two-week Treatment phase (Days 15-28), Four-week Post-treatment phase (Days 29-56)
  On each study day, participants will receive EMA text surveys on their cellphones. For each participant, cannabis use frequency will be measured as the number of days per week they report cannabis use. During the two-week pre-treatment period, we will calculate the baseline frequency as the average number of use days per week across those two weeks. Cannabis use frequency will then be assessed during each of the two treatment weeks (Week 0-1) and during the four-week follow-up period (Weeks 2-5), and the follow-up period will subsequently be compared relative to baseline. This is corroborated by TLFB.
Quantity of cannabis use | Two-week Pre-treatment/Baseline phase (Days 1-14), Two-week Treatment phase (Days 15-28), Four-week Post-treatment phase (Days 29-56)
  On each study day, participants will receive EMA text surveys on their cellphones. For each participant, cannabis use quantity will be measured as the average number of grams used per use-day during each week in which they report cannabis use. During the two-week pre-treatment/baseline period (Days 1-14), we will calculate the baseline quantity as the average daily grams used per use-day across those two weeks. Cannabis use quantity will then be assessed during the treatment phase (Days 15-28) and during the 4-week follow-up period (Days 29-56), and the follow-up period will subsequently be compared relative to baseline. This will be corroborated by TLFB.

SECONDARY OUTCOMES:
Salience Network drug cue reactivity | Pre-treatment/Baseline (Day 14), Immediate Post-treatment (Day 28), 4-Week Post-treatment Follow-up (Day 56)
  Brain activity in response to cannabis-related versus neutral cues will be assessed using the Cannabis Stroop fMRI task, in which visual stimuli are presented and the Salience Network (SN) typically shows greater activation to drug cues than to neutral cues. This pattern reflects heightened SN drug-cue reactivity, or an attentional bias toward drug-related information. First, a data-driven approach called independent component analysis (ICA) will be used to identify and extract the SN timecourse and spatial map from the Stroop fMRI task data. Second, a general linear model (GLM) analysis will be used to relate each participant's SN timecourse to the task design (timing model of cue presentation blocks), allowing us to quantify SN activity during cannabis versus neutral cue task conditions. The primary outcome will be each participant's SN contrast beta value, a statistic derived from the ICA-GLM analysis that reflects the magnitude and direction of SN drug cue reactivity.
Feasibility (attendance) | Two-week Treatment phase (Days 15-28)
  Feasibility will be measured as the percentage of scheduled TMS sessions completed by participants in each treatment group. For participants randomized to a TMS treatment group (active vs. sham) who attend at least one TMS session, we will quantify the total number of sessions completed. Feasibility will then be calculated as the percentage of planned TMS sessions that were successfully completed by each participant.
Tolerability (withdrawals) | Two-week Treatment phase (Days 15-28)
  Tolerability will be measured as the proportion of participants who withdraw from the study before completing all planned TMS sessions. Among participants randomized to a TMS treatment group (active vs. sham) who attend at least one TMS session, we will identify those who discontinue prior to completing their final scheduled TMS session. Tolerability will then be quantified as the percentage of participants who withdraw before completing the full course of planned TMS treatments.
Safety (AEs) | Two-week Treatment phase (Days 15-28)
  Safety will be measured as the frequency, type, and severity of treatment-related adverse events (AEs) reported during and after the TMS treatment period, categorized according to standard AE reporting guidelines. Among participants randomized to a TMS treatment group (active vs. sham) who attend at least one TMS session and receive any amount of TMS, we will quantify the number, type, and severity of subsequent treatment-related AEs. Adverse event profiles will then be compared between the active and sham treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Tonisha Kearney-Ramos, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No